CLINICAL TRIAL: NCT02603029
Title: Placebo Controlled Study of Influence of Cream With the Silver Fir (Abies Alba) Wood Extract on the Skin
Brief Title: Influence of of Cream With the Silver Fir Wood Extract (Belinal) on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Abies Labs d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Belinal 01-2015
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2015-11

CONDITIONS: Wrinkles; Ageing; Photoprotection; Skin Care; Skin Cream
Keywords: skin rejuvenation; anti-ageing effects; minimal erythema dose; dermis structure; physiological skin condition; wrinkling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo cream (Placebo Comparator): Cream with 0% Silver fir wood extract (Belinal)
  Interventions: Other: Placebo cream
- Belinal cream (Active Comparator): Cream with 2% Silver fir wood extract (Belinal)
  Interventions: Other: Belinal cream

INTERVENTIONS:
Other: Placebo cream — Subjects will use placebo cream twice per day for 12 weeks on one half of the face and of the gluteal area.
  Arms: Placebo cream
Other: Belinal cream — Subjects will use Belinal cream twice per day for 12 weeks on the other half of the face and of the gluteal area.
  Arms: Belinal cream

SUMMARY:
Objective of the study is to determine the influence of the cream with Silver fir wood (Abies alba) extract (Belinal) on the skin parameters and functions in comparison to the placebo cream. 10 healthy female subjects will use the test cream on one half and placebo cream on the other half of the face and of the gluteal part twice a day for 12 weeks. Various face skin parameters will be evaluated before the cream use (the baseline), after 6 and after 12 weeks of the cream use. To evaluate the photoprotective potential of Belinal the minimal erythema dose (MED) will be determined before (the baseline) and after 12 weeks of the cream use at the gluteal area.

DETAILED DESCRIPTION:
Objective of the study is to determine the influence of the cream with Silver fir wood (Abies alba) extract (Belinal; 2% cream) on the skin parameters and functions in comparison to the placebo cream. 10 healthy female subjects will use the test cream on one half and placebo cream on the other half of the face and of the gluteal area (split-face and split-gluteal area ) twice a day for 12 weeks. Face skin parameters will be evaluated before the cream use (the baseline), after 6 and after 12 weeks of the cream use. The photoprotective potential of Belinal will be evaluated with a determination of the minimal erythema dose (MED) at the gluteal area before (the baseline) and after 12 weeks of the cream use. Comparison will be done as the mean of the individual ratios. The differences between the before-after condition will be analyzed with the statistical test of analysis of variance. In case of failure to find homogeneity in the variances the nonparametric ANOVA, the Willcoxon test, will be used. The results will be expressed as mean ± standard error for each group with a significance level of 0.05 for all the statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Signs of skin aging (mimic wrinkles/ fine lines/ poor skin tone/ photoaged skin),
* Phototype II and III.

Exclusion Criteria:

* Allergy to ingredients of tested products
* Diagnosed diabetes
* Thyroid disease
* Inflammatory dermatoses
* Regular use of dietary supplements 6 months or less before start of the study,
* Invasive rejuvenation treatments (botox injections, hyaluronic acid fillers, needle rollers, needle mesotherapy, etc.) 6 months or less prior to start of the study,
* Non-invasive rejuvenation treatments (radiofrequency, electrotherapy, ultrasound therapy, no-needle mesotherapy, etc.) 3 months or less prior to start of the study,
* Regular, at least 14 day use of anti-aging cosmetic products containing peptides/ polyphenols/ stem cells extracts/ vitamins in high concentration/ AHAs/ BHAs/ vitamin A or its derivatives) three months or less prior to start of the study,
* Gluteal hyperpigmentation,
* Expected sunbathing (also in solariums) within the study period.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Improvement of photoprotective function of the skin | up to 12 weeks of the supplementation
  Minimal erythema dose (MED) of the skin will be determined. Skin on the gluteal part of the body will be exposed to 10 different doses of UVB light and 24 hours after exposure MED will be determined. Higher MED indicates better photoprotective function of the skin.
Improvement of the dermis structure | up to 12 weeks of Belinal cream use
  Ultrasound (US) images of the dermis will be taken and intensity of the dermis determined. Higher intensity of the dermis US images indicates improvement of the collagen and elastin network.

SECONDARY OUTCOMES:
Reduction of the area of the periorbital facial wrinkles | 6 and 12 weeks of Belinal cream use
  Area of selected periorbital wrinkles will be quantitatively assessed using CSI programme.
Reduction of the volume of the periorbital facial wrinkles | 6 and 12 weeks of Belinal cream use
  Volume of selected periorbital wrinkles will be quantitatively assessed using CSI programme.
Reduction of trans-epidermal water loss | 6 and 12 weeks of Belinal cream use
  Trans-epidermal water loss (TEWL) will be measured on the face using open-chamber probe. Lower TEWL indicates better skin barrier function and improved skin condition.
Improved skin hydration | 6 and 12 weeks of Belinal cream use
  Skin hydration will be measured on the face.
Improved skin elasticity | 6 and 12 weeks of Belinal cream use
  Skin elasticity will be measured on the face.
An increase of the dermis thickness | 6 and 12 weeks of Belinal cream use
  Dermis thickness will be measured with ultrasound imaging of the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Janko Zmitek, PhD, Study Chair — VIST - Faculty of Applied Sciences; Katja Zmitek, PhD, Study Director — VIST - Faculty of Applied Sciences; Nataša Tavčar, BSc, Principal Investigator — VIST - Faculty of Applied Sciences; Tina Pogačnik, BSc, Principal Investigator — VIST - Faculty of Applied Sciences